CLINICAL TRIAL: NCT02466568
Title: A Randomized Phase I/II Study of Nivolumab in Combination With GM.CD40L Vaccine in Adenocarcinoma of the Lung
Brief Title: Study of Nivolumab in Combination With GM.CD40L Vaccine in Adenocarcinoma of the Lung
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18147; 1504-1392 (Other: NIH Office of Biotechnology Activities (OBA))
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer; Adenocarcinoma of the Lung
Keywords: advanced; metastatic; lung disease; adenocarcinoma; non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Neoplasm Metastasis; Lung Diseases; Adenocarcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; spartalizumab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I and Phase II Treatment Arm (Experimental): Participants will receive nivolumab and GM.CD40L. Treatment will be administered on an outpatient basis. The nivolumab will be given first followed by the GM.CD40L vaccine for those enrolled on this arm.
  Interventions: Drug: Nivolumab; Biological: GM.CD40L Vaccine
- Phase II Control Arm (Active Comparator): Nivolumab treatment without GM.CD40L. Nivolumab will be given every 2 weeks at a dose of 3mg/kg.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Participants will receive treatment with nivolumab as a 60-minute +/-5 minutes intravenous (IV) infusion on Day 1 and 15 of each 28-day cycle.
  Other Names: Opdivo; Anti-PD-1
Biological: GM.CD40L Vaccine — GM.CD40L will be injected intradermally every 2 weeks for 4 injections, then every month for 4 injections, then every 3 months until the patient is off treatment.
  Other Names: Immunotherapy; Cell Vaccine
  Arms: Phase I and Phase II Treatment Arm

SUMMARY:
The purpose of this study is to find out what effects (good and bad) a tumor vaccine (GM.CD40L) used in combination with Nivolumab will have on participants and their cancer. Another purpose of the study is to find out the maximum tolerated dose of nivolumab in combination with GM.CD40L vaccine. Investigators also want to find out if the combination of GM.CD40L and nivolumab can boost the immune system of participants like you, and how their immune system reacts, both before and after the treatment.

DETAILED DESCRIPTION:
This study has two parts and participants may be involved in either Phase I part or Phase II.

Phase I: Investigators plan to enroll participants in cohorts of 6 and monitor side effects over a 21 day period to determine the maximum tolerated dose (MTD) of nivolumab, which will be given in combination with GM.CD40L. This is being done since this study involves a combination of treatments that have not been studied in humans before and to find the best dose for the Phase II part of the study.

Phase II: Investigators plan to compare any clinical benefit in the participants who receive the combination of GM.CD40L vaccine with nivolumab, to participants that receive only nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of advanced/metastatic adenocarcinoma of the lung
* Eastern Cooperative Oncology Group (ECOG) performance status of 0/1
* Chemotherapy naïve or have completed adjuvant chemotherapy for non-small cell lung cancer (NSCLC) >6 months prior
* Adequate bone marrow, renal and hepatic function
* Must have measurable metastatic disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
* Mandatory archival tissue or willingness to undergo a fresh biopsy
* Life expectancy of greater than 6 months

Exclusion Criteria:

* Symptomatic brain metastasis or uncontrolled central nervous system (CNS) metastasis
* Pregnancy or breast feeding
* Serious uncontrolled medical disorder or active infection that would impair the participant's ability to receive study treatment
* Prior use of a PD1 or PDL1 inhibitor
* Concurrent use of other anticancer approved or investigational agents is not allowed
* Autoimmune disorders
* Prior malignancy in past 2 years
* Systemic steroids at doses greater than 10 mg/day of prednisone or the equivalent
* Any other pre-existing immunodeficiency condition (including known HIV infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Phase I: Recommended Phase II Dose | Up to 2 months
  The recommended Phase II dose will be defined as the highest dose level of GMCD40L vaccine in combination with nivolumab that induced dose limiting toxicity (DLT) in fewer than 33% of patients.
Phase II: Objective Response Rate (ORR) | Up to 2 years
  Objective tumor response per treatment arm. ORR: Complete Response (CR) = disappearance of all target lesions + Partial Response (PR) = 30% decrease in the sum of the longest diameter of target lesions.

SECONDARY OUTCOMES:
Phase II: Overall Survival (OS) | Up to 2 years
  OS per treatment arm. Overall survival is defined as the time from randomization until death from any cause.
Phase II: Progression-free Survival (PFS) | Up to 2 years
  PFS per treatment arm. Progressive Disease (PD): = 20% increase in the sum of the longest diameter of target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Jhanelle Gray, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute